CLINICAL TRIAL: NCT05445856
Title: Intraoperative Methadone for Postoperative Pain in Patients Undergoing Tonsillectomy - a Randomized Controlled Trial
Brief Title: Intraoperative Methadone for Postoperative Pain in Patients Undergoing Tonsillectomy
Acronym: METATONS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-002496-11
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Methadone
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone (Experimental): Single-shot intravenous methadone 0.2 mg/kg administered intraoperatively
  Interventions: Drug: Methadone
- Fentanyl (Active Comparator): Single-shot intravenous fentanyl 3 microgram/kg administered intraoperatively
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Methadone — Methadone is administered as a single intravenous dose after induction of anesthesia and prior to initiation of surgery
  Arms: Methadone
Drug: Fentanyl — Fentanyl is administered as a single intravenous dose after induction of anesthesia and prior to initiation of surgery
  Arms: Fentanyl

SUMMARY:
A randomized controlled trial evaluating the efficacy and safety of single-shot intraoperative methadone for postoperative pain in patients undergoing tonsillectomy. Fentanyl is used as an active comparator

DETAILED DESCRIPTION:
This study is an investigator-initiated, prospective, randomised controlled trial with two arms: an intervention arm (methadone) and a control arm (fentanyl). Patients scheduled for tonsillectomy at Randers Regional Hospital, Denmark, will be approached for study participation.

Patients are randomised in a 1:1 ratio in blocks of varying sizes (between 4 and 8) to receive either intraoperative methadone or fentanyl. The randomisation assignment will be handled by the hospital pharmacy using a web-based central randomisation procedure (www.sealedenvelope.com).

The study drug will be prepared by the hospital pharmacy at Aarhus University Hospital and delivered as kits with identical appearance, marked with the randomization number (1-130). On the day of surgery, a kit will be opened and a 10 ml syringe with study drug (methadone 2 mg/ml or fentanyl 30 microgram/ml or ) will prepared by a health care professional (nurse or medical doctor not involved in the study or the treatment of patients). Once prepared, the blinded study drug will be given to and handled by one of the research team members and administered after induction of anesthesia and prior to surgery

The dose of the study drug will be administered as intravenous bolus dose in equipotent doses (0.2 mg/kg / 3 μg/kg) corresponding to 1 ml for every 10 kg of ideal body weight (women: height (cm) - 105. Men: height (cm) - 100)) after induction of anaesthesia and before the start of surgery.

Postoperative data will be obtained by reviewing hospital records, by interview and electronic questionnaires sent by email.

ELIGIBILITY:
Inclusion Criteria:

* All patients (≥18 years) scheduled for elective tonsillectomy

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status IV or V
* Allergy to study drugs
* Daily use of opioids 7 days prior to surgery
* Inability to provide informed consent
* Severe respiratory insufficiency
* Heart failure
* Acute alcohol intoxication/delirium tremens
* Increased intracranial pressure
* Acute liver disease
* Liver insufficiency
* Kidney insufficiency
* Treatment with rifampicin
* Treatment with any drug prolonging the QT-interval
* Pregnancy (every female not using contraceptives will be screened with urine human choriogonadotropin)
* Breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | On arrival at the post-anesthesia care unit
  Pain at swallowing (numeric rating scale (NRS) 0-10, lower scores are better outcomes)
Opioid consumption | First 5 postoperative days
  Cumulative postoperative opioid consumption in morphine equivalents

SECONDARY OUTCOMES:
Postoperative pain | 1, 2, 3, 5 and 7 days after surgery
  Pain at swallowing (numeric rating scale (NRS) 0-10, lower scores are better outcomes)
Opioid consumption | 1 and 7 days after surgery
  Cumulative postoperative opioid consumption in morphine equivalents
Postoperative nausea and vomiting (none, mild, moderate, severe) | 1, 2 and 3 days after surgery
  Nausea and/or vomiting (PONV), proportion of patients with none or mild PONV
Sedation | 4 hours after surgery
  Level of sedation (Ramsay Scale (1-4)), proportion of patients being co-operative, oriented and tranquil

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, PhD, DMSc, Study Chair — Aarhus University Hospital, Department of Anesthesia and Intensive Care
Locations (1):
- Department of Anaesthesiology and Intensive Care, Randers, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request

REFERENCES:
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Vender JS, Benson J, Newmark RL. Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Posterior Spinal Fusion Surgery: A Randomized, Double-blinded, Controlled Trial. Anesthesiology. 2017 May;126(5):822-833. doi: 10.1097/ALN.0000000000001609. PMID 28418966
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Udelsmann A, Maciel FG, Servian DC, Reis E, de Azevedo TM, Melo Mde S. Methadone and morphine during anesthesia induction for cardiac surgery. Repercussion in postoperative analgesia and prevalence of nausea and vomiting. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):695-701. doi: 10.1016/S0034-7094(11)70078-2. English, Multiple languages. PMID 22063370
- [Derived] Bondergaard M, Uhrbrand PG, Karaca T, Rhode M, Kjaergaard T, Svendsen RT, Klug TE, Nikolajsen L, Friesgaard KD. Intraoperative methadone for postoperative pain in adult patients undergoing tonsillectomy-a randomised controlled trial. BJA Open. 2025 May 26;14:100418. doi: 10.1016/j.bjao.2025.100418. eCollection 2025 Jun. PMID 40502985